CLINICAL TRIAL: NCT04722588
Title: Integrating the Clinical Pharmacist Into the Emergency Department Interdisciplinary Team: A Study Protocol for a Multicentre Trial Applying a Non-randomized Stepped Wedge Study Design
Brief Title: Integrating the Clinical Pharmacists Into Emergency Department Teams
Acronym: ED-PHARM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Pharmacy of North Norway Trust (Other)
Collaborators: University Hospital of North Norway (Other); Nordlandssykehuset HF (Other); The Royal Norwegian Ministry of Health (Other); University of Tromso (Other)
Responsible Party: Principal Investigator, Renate Elenjord, Philosophia Doctor, Hospital Pharmacy of North Norway Trust
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HPNorhNorway
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Emergency Department; Clinical Pharmacist
Keywords: Medication therapy; Clinical pharmacist; Interdisciplinary team collaboration; Emergency department; Stepped-wedge trial
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: The intervention comprises implementing the clinical pharmacists in the interdisciplinary team in three emergency departments (EDs) in Northern Norway. A non-randomized stepped-wedge design will be applied. This design allows the intervention to be rolled out sequential, allowing us to control for differences between study sites (vertical control) and secular trends (horizontal control) during the study period. This is the gold standard when a conventional randomized controlled trial is not possible.
  The intervention will be implemented over a 12-month period, starting with a three-month control period in all EDs. This period allows for baseline data collection before the intervention. After this period, the investigators will consecutively roll out the intervention at three months interval to the EDs. The intervention will start in Tromsø, which is the largest ED, continue in Bodø and finish in Harstad, which is the smallest of the three EDs.
Masking Description: Masking members of the interdisciplinary team is not possible as a new member of staff is being introduced. However, the study will not be announced to patients presenting to the EDs.
  Patients will know that there is a study ongoing, but will not have to consent to participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control period (No Intervention): The control period is represented by standard care procedures, which are similar in all three EDs: Patients cared for in the EDs receive treatment from ED physicians and nurses, and no pharmacists are involved in any of the EDs.
- Intervention period (Experimental): During the intervention period, clinical pharmacists will be present in the EDs from 08.00 - 19.00 Monday to Friday.
  The ED pharmacists will collaborate with the interdisciplinary team and perform the following tasks as appropriately as possible and by prioritized need; medication history taking, medication reconciliation, medication review, drug therapy recommendations, guidance on drug administration, medication information and counseling to patients/next of kin and health care personnel and communication about medications and changes in medication regimes. Standardized procedures, like the integrated medicines management (IMM) methodology, will be applied where possible. How, when and which task will be performed for each patient cannot be predetermined, but must be performed according to patient's needs and eventual time constraints.
  Interventions: Other: Introducing clinical pharmacists to the interdisciplinary ED team.

INTERVENTIONS:
Other: Introducing clinical pharmacists to the interdisciplinary ED team. — There will be two shifts, one shift from 08.00 - 15.00 and one from 12.00 - 19.00. Consequently, the hours of the day when the majority of patients arrives, are covered and the pharmacist capacity is doubled during the busiest time of the day. Early mornings are normally relatively slowed paced and the pharmacist may use this time to follow up on patients admitted during the night (from 19.00 - 08.00), in particularly those who have been admitted to wards without an assigned pharmacist.
  Arms: Intervention period

SUMMARY:
The "Emergency Department (ED) Pharmacist" is an integrated part of the ED interdisciplinary team in many countries, which have shown to improve medication safety and reduce costs related to hospitalisations. In Norway, few EDs are equipped with an ED pharmacist, and research describing effects on patients has not been conducted.

This is a multicentre study where the intervention will be implemented in the regular operation of three EDs in Northern Norway; Tromsø, Bodø and Harstad.

Clinical pharmacists will work as an integrated part of the ED team, and provide pharmaceutical care services such as medication reconciliation, medication review or medication counselling. The medical condition and complexity of the patient's disease will influence the extend and type of service from the pharmacist.

A non-randomized stepped wedge study design will be applied, where the ED pharmacist will be implemented in all three EDs after a three, six- and nine- month control period, respectively. Each ED will consequently have both intervention and control periods.

All patients going through the three EDs during the 12-month study period will be included. Patients admitted in the control periods will be allocated to the control group, while patients admitted in the intervention periods will be allocated to the intervention group.

The primary endpoint is "Time in hospital during 30 days after admission to the ED", which is a composite endpoint combining i) time in ED during stay, ii) time in hospital during stay if hospitalized and iii) time in urgent care clinic, ED and/or hospital if rehospitalized within 30 days after admission to ED Secondary endpoints include time to rehospitalization, length of stay (LOS) during first hospitalisation, LOS in EDs, rehospitalisation rates and mortality rates.

Patient data will be collected retrospectively from national data registries, from the hospital system and from patient records.

The Regional Committee for Medical and Health Research Ethics and Local Patient Protection Officers in all hospitals have approved the study.

DETAILED DESCRIPTION:
The intervention will be assessed using a non-randomized stepped wedge trial design. A stepped wedge design allows for the intervention to be rolled out at different times, thus allowing us to control for differences between study sites (vertical control) and secular trends (horizontal control) during the study period. This is the gold standard when a conventional randomized controlled trial is not possible.

The stepped wedge study design is based on a staggered implementation of the intervention in the intervention sites. This will be done over a 12-month period, starting with a three-month control period in all EDs (planned start-up February 1st, 2021). This period allows for baseline data collection before the intervention. After this period, the investigators will consecutively roll out the intervention at three months interval to the EDs. The intervention will start in Tromsø which is the largest ED, continue in Bodø and finish in Harstad, which is the smallest of the three EDs. After nine months, all EDs will have clinical pharmacists. When the intervention is implemented in an ED, it will continue until the trial is terminated (planned January 31th, 2022).

This is a multicentre study including three EDs in Northern Norway Health Authority region; the University Hospital of North Norway (UNN) Tromsø, Nordland Hospital (NLSH) in Bodø and UNN Harstad with approximately 15 000, 12 000 and 6000 patients presenting annually in the respective EDs. These numbers include patients being admitted more than once to the ED. The three EDs operate similarly and receive patients who need immediate health care in case of acute illness or injury. Norway has a well-functioning primary care system, including municipal urgent care clinics providing ambulatory care outside of general practitioner (GP) office hours. In order to be admitted to the ED, the patients need a referral either from GP or from a physician at an urgent care clinic. At the ED, the patient is met by an ED nurse and an ED physician (either an intern or a resident in specialty training), who perform the initial examinations and assessments of the patient. A senior physician is always on call in case of the need for a consultation. NLSH is the only ED with senior physicians situated in the ED during day-time. From the ED, patients are either admitted to a hospital ward, transferred to a municipally run health institution or discharged to their homes.

All patients presenting to the EDs during the study period will be included. Patients presenting during the control period, will be allocated to the control group (n≈14400), while patients presenting during the intervention period will be allocated to the intervention group (n≈19200), independently of whether they receive clinical pharmacist services or not. Patients for whom data is not available retrospectively, will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to the EDs during the study period will be included.

Exclusion Criteria:

* Patients for whom data is not available retrospectively.
* Patients who actively ask not to be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30888 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time in hospital during 30 days after admission to the ED | 30 days
  This is a composite endpoint adding times during a 30-day period accounted from admission in ED for the first time in trial period (index stay): 1) time in ED during index stay, 2) time in hospital during index stay if hospitalized and 3) time in ED or hospital if rehospitalized within 30 days after index admission to ED.

SECONDARY OUTCOMES:
Time to rehospitalization (unplanned) or visit to urgent care clinic | 30 days
  Time before the first unplanned rehospitalization or visit to urgent care clinic will be measured and the duration from the control period to the duration from the intervention period will be compared.
30-day rate for rehospitalization or visit to urgent care clinic (unplanned) | 30 days
  The 30-day rate for rehospitalization or visit to urgent care clinic during the control period will be compared with the trial period where an ED pharmacist will be present in the ED. The rate will be measured by the number of patients who are rehospitalized within 30 days after their stay.
Length of stay in hospital | 30 days
  Length of stay (LOS) in hospital will be calculated as discharge date minus admission date. The LOS in hospital for all patients in the trial period in all three EDs will be calculated.
Length of stay in ED | 48 hours
  The ED LOS will be represented in minutes as discharge time from the ED (or time transferred to a hospital ward) minus admission time in the ED.
Mortality ratio | 30 days
  The proportion of patients who died within 30 days of admission to the ED in the control period compared to the intervention period.
Time to death | 30 days
  Number of days from admission to the ED until death will be measured and compared between control and intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Renate Elenjord, PhD, Principal Investigator — Hospital Pharmacy of North Norway Trust
Locations (3):
- Norway (3):
  - Nordlandssykehuset HF, Bodø
  - University hospital of north norway, Harstad
  - University hospital of North Norway, Tromsø

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vesela R, Elenjord R, Lehnbom EC, Ofstad EH, Johnsgard T, Zahl-Holmstad B, Risor T, Wisloff T, Roslie L, Filseth OM, Valle PC, Svendsen K, Froyshov HM, Garcia BH. Integrating the clinical pharmacist into the emergency department interdisciplinary team: a study protocol for a multicentre trial applying a non-randomised stepped-wedge study design. BMJ Open. 2021 Nov 25;11(11):e049645. doi: 10.1136/bmjopen-2021-049645. PMID 34824109